CLINICAL TRIAL: NCT03451890
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of E2730 in Healthy Subjects
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of E2730 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2730-A001-002
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2018-02

CONDITIONS: Healthy Participants
Keywords: Healthy participants; E2730; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1: E2730 40 mg (Experimental): Participants will receive a single oral dose of E2730 40 milligrams (mg) under fasted conditions.
  Interventions: Drug: E2730
- Cohort 1: Matching placebo (Placebo Comparator): Participants will receive a single oral dose of matching placebo under fasted conditions.
  Interventions: Drug: Placebo
- Cohort 2: E2730 80 mg (Experimental): Participants will receive a single oral dose of E2730 80 mg under fasted conditions.
  Interventions: Drug: E2730
- Cohort 2: Matching placebo (Placebo Comparator): Participants will receive a single oral dose of matching placebo under fasted conditions.
  Interventions: Drug: Placebo
- Cohort 3: E2730 120 mg (Experimental): Participants will receive a single oral dose of E2730 120 mg under fasted conditions.
  Interventions: Drug: E2730
- Cohort 3: Matching placebo (Placebo Comparator): Participants will receive a single oral dose of matching placebo under fasted conditions.
  Interventions: Drug: Placebo
- Cohort 4: E2730 160 mg (Experimental): Participants will receive a single oral dose of E2730 160 mg under fasted conditions.
  Interventions: Drug: E2730
- Cohort 4: Matching placebo (Placebo Comparator): Participants will receive a single oral dose of matching placebo under fasted conditions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E2730 — oral capsule
  Arms: Cohort 1: E2730 40 mg; Cohort 2: E2730 80 mg; Cohort 3: E2730 120 mg; Cohort 4: E2730 160 mg
Drug: Placebo — oral capsule
  Arms: Cohort 1: Matching placebo; Cohort 2: Matching placebo; Cohort 3: Matching placebo; Cohort 4: Matching placebo

SUMMARY:
This study will be conducted to evaluate the safety, tolerability, and pharmacokinetics of single ascending oral doses of E2730 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, male or female, age ≥18 years and ≤55 years old at the time of informed consent (Note: To be considered non-smokers, participants must have discontinued smoking for at least 4 weeks before dosing.)
* Body mass index (BMI) ≥18 and <32 kilograms per meters squared (kg/m^2) at Screening

Exclusion Criteria:

* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [β-hCG] or human chorionic gonadotropin [hCG] test with a minimum sensitivity of 25 International Units per liter (IU/L) or equivalent units of β-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
* Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period or for 5 times the half-life of the study drug plus 90 days after study drug discontinuation). No sperm donation is allowed during the study period and for 5 times the half-life of the study drug plus 90 days after study drug discontinuation.
* Participants with history of seizures, including those experienced in childhood
* Any history of gastrointestinal surgery that may affect pharmacokinetic profiles of E2730, e.g., hepatectomy, nephrectomy, and digestive organ resection
* A prolonged QT/QTc interval (QTcF >450 milliseconds) demonstrated by a repeated ECG at Screening or Baseline (based on average of triplicate ECGs). A history of risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of long QT Syndrome) or the use of concomitant medications that prolonged the QT/QTc interval
* Persistent systolic blood pressure (BP) >139 or <90 millimeters of mercury (mmHg) or diastolic BP >89 or <50 mmHg at Screening or Baseline
* Left bundle branch block
* History of myocardial infarction or active ischemic heart disease
* History of clinically significant arrhythmia or uncontrolled arrhythmia
* Known history of clinically significant drug allergy at Screening
* Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening
* Known to be human immunodeficiency virus (HIV) positive at Screening
* Active viral hepatitis (A, B, or C) as demonstrated by positive serology at Screening
* History of drug or alcohol dependency or abuse, or those who have a positive drug test at Screening or Baseline
* Currently enrolled in another clinical study or used any investigational drug or device within 28 days or 5 half-lives, whichever is longer, preceding informed consent
* Participants who undergo blood transfusion within 12 weeks, or who donate 400 milliliters (mL) or more of whole blood within 12 weeks or 200 mL or more of whole blood within 4 weeks, or who make a component donation within 2 weeks prior to dosing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Mean maximum observed concentration (Cmax) for E2730 and the N-acetyl metabolite (M1) in plasma | predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, and 12 hours (hr) postdose (PD) on Day 1; thereafter on Day 2 (24 hr PD), Day 3 (48 hr PD), Day 4 (72 hr PD), Day 5 (96 hr PD), Day 6 (120 hr PD), Day 7 (144 hr PD), and Day 10 (216 hr PD), and Day 13 (288 hr PD)
Time at which the highest drug concentration (tmax) occurs for E2730 and the N-acetyl metabolite (M1) in plasma | predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, and 12 hours (hr) postdose (PD) on Day 1; thereafter on Day 2 (24 hr PD), Day 3 (48 hr PD), Day 4 (72 hr PD), Day 5 (96 hr PD), Day 6 (120 hr PD), Day 7 (144 hr PD), and Day 10 (216 hr PD), and Day 13 (288 hr PD)
Mean area under the concentration-time curve from zero time to 24 hours after dosing (AUC[0-24h]) for E2730 and the N-acetyl metabolite (M1) in plasma | predose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, and 12 hours postdose on Day 1; Day 2 (24 hours postdose)
Mean area under the concentration-time curve from zero time to time of last quantifiable concentration (AUC[0-t]) for E2730 and the N-acetyl metabolite (M1) in plasma | predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, and 12 hours (hr) postdose (PD) on Day 1; thereafter on Day 2 (24 hr PD), Day 3 (48 hr PD), Day 4 (72 hr PD), Day 5 (96 hr PD), Day 6 (120 hr PD), Day 7 (144 hr PD), and Day 10 (216 hr PD), and Day 13 (288 hr PD)
Mean area under the concentration-time curve from zero time to 72 hours after dosing (AUC[0-72h]) for E2730 and the N-acetyl metabolite (M1) in plasma | predose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, and 12 hours postdose on Day 1; thereafter on Day 2 (24 hours postdose), Day 3 (48 hours postdose), Day 4 (72 hours postdose)
Mean area under the concentration-time curve from zero time extrapolated to infinite time (AUC[0-inf]) for E2730 and the N-acetyl metabolite (M1) in plasma | predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, and 12 hours (hr) postdose (PD) on Day 1; thereafter on Day 2 (24 hr PD), Day 3 (48 hr PD), Day 4 (72 hr PD), Day 5 (96 hr PD), Day 6 (120 hr PD), Day 7 (144 hr PD), and Day 10 (216 hr PD), and Day 13 (288 hr PD)
Mean terminal elimination phase half-life (t1/2) for E2730 and the N-acetyl metabolite (M1) in plasma | predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, and 12 hours (hr) postdose (PD) on Day 1; thereafter on Day 2 (24 hr PD), Day 3 (48 hr PD), Day 4 (72 hr PD), Day 5 (96 hr PD), Day 6 (120 hr PD), Day 7 (144 hr PD), and Day 10 (216 hr PD), and Day 13 (288 hr PD)
Mean apparent total clearance following oral administration (CL/F) of E2730 | predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, and 12 hours (hr) postdose (PD) on Day 1; thereafter on Day 2 (24 hr PD), Day 3 (48 hr PD), Day 4 (72 hr PD), Day 5 (96 hr PD), Day 6 (120 hr PD), Day 7 (144 hr PD), and Day 10 (216 hr PD), and Day 13 (288 hr PD)
Mean apparent volume of distribution at terminal phase (Vz/F) for E2730 in plasma | predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, and 12 hours (hr) postdose (PD) on Day 1; thereafter on Day 2 (24 hr PD), Day 3 (48 hr PD), Day 4 (72 hr PD), Day 5 (96 hr PD), Day 6 (120 hr PD), Day 7 (144 hr PD), Day 10 (216 hr PD), and Day 13 (288 hr PD)
Mean metabolite ratio (%) (MRP) in plasma | predose; 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, and 12 hours (hr) postdose (PD) on Day 1; thereafter on Day 2 (24 hr PD), Day 3 (48 hr PD), Day 4 (72 hr PD), Day 5 (96 hr PD), Day 6 (120 hr PD), Day 7 (144 hr PD), and Day 10 (216 hr PD), and Day 13 (288 hr PD)
  Metabolite ratio (%) is calculated as the ratio of plasma AUC(0-inf) of a metabolite to a parent following molar correction.
Mean amount of unchanged drug excreted (Ae) in urine for E2730 and the N-acetyl metabolite (M1) | Days 1 through Days 7 at the following intervals: predose; 0 to 4, >4 to 8, >8 to 12, >12 to 24, >24 to 48, >48 to 72, >72 to 96, >96 to 120, and >120 to 144 hours postdose
Renal clearance (CLR) of E2730 and the N-acetyl metabolite (M1) | Days 1 through Days 7 at the following intervals: predose; 0 to 4, >4 to 8, >8 to 12, >12 to 24, >24 to 48, >48 to 72, >72 to 96, >96 to 120, and >120 to 144 hours postdose
Percent (%) of administered dose of E2730 and the N-acetyl metabolite (M1) excreted in urine | Days 1 through Days 7 at the following intervals: predose; 0 to 4, >4 to 8, >8 to 12, >12 to 24, >24 to 48, >48 to 72, >72 to 96, >96 to 120, and >120 to 144 hours postdose
Mean metabolite ratio (%) (MRP) for E2730 and the N-acetyl metabolite (M1) in urine | Days 1 through Days 7 at the following intervals: predose; 0 to 4, >4 to 8, >8 to 12, >12 to 24, >24 to 48, >48 to 72, >72 to 96, >96 to 120, and >120 to 144 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Collaborative Neuroscience Network, Long Beach, California, United States